CLINICAL TRIAL: NCT01324843
Title: Safety and Tolerability of the Derma Vax Clinical Intradermal Electroporation System in Healthy Subjects
Brief Title: Safety and Tolerability of the Derma Vax(Trademark) Clinical Intradermal Electroporation System in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 999909249; 09-AG-N249
Record Dates: First submitted 2011-03-26; First posted 2011-03-29 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-09-20

CONDITIONS: Intradermal Electroporation
Keywords: Safety and Tolerability; Intradermal Electroporation
MeSH Terms: interventions — Lidocaine, Prilocaine Drug Combination

INTERVENTIONS:
Drug: EMLA Cream
Drug: Aveeno Daily Moist
Device: Derma Vax
Procedure: Intradermal Electroporation
Procedure: Visual Analogue Scale
Procedure: Present Pain Intensity
Procedure: McGill Pain Questionnaire
Procedure: Skin Assessment

SUMMARY:
Background:

- Researchers are investigating the use of DNA vaccines to treat various types of cancer by provoking an immune system response to tumor cells. DNA vaccines mimic the effect of normal vaccines given to prevent infectious diseases, but they have been less effective than anticipated in humans. To improve the effectiveness of DNA vaccines, researchers are studying alternate delivery methods, such as the investigational Derma Vax(Trademark) injection system that delivers the vaccine into the skin. However, because the Derma Vax(Trademark) system has not been studied in humans, more research is needed to determine whether this new vaccine delivery method is safe and tolerable, particularly in terms of pain levels and skin reactions.

Objectives:

- To evaluate the safety, effectiveness, and relative pain levels of intradermal electroporation using Derma Vax(Trademark) administered after pretreatment with either a topical cream anesthetic or placebo cream.

Eligibility:

- Healthy individuals between 18 and 55 years of age.

Design:

* Participants will be screened with a medical history, physical examination, blood and urine tests, and an electrocardiogram.
* Participants will have two different creams applied to their upper arms: one cream will be an anesthetic (lidocaine and prilocaine) and the other will be a placebo lotion. Each arm will receive a different cream.
* Once the cream has taken effect, participants will receive Derma Vax(Trademark) treatment. No actual medication will be given during the injection; participants will evaluate their reaction based on the pressure and needle stick alone.
* Immediately after the treatment, participants will use the Visual Analogue Scale of pain intensity to provide a description of the level of pain experienced during the injection.
* Participants will complete additional questionnaires about pain intensity and will have the injected skin site inspected to determine possible reactions to the injection. They will also be asked their opinions on whether (based on pain levels) a series of Derma Vax(Trademark) treatments would be acceptable for treatment of a serious illness.
* The day after the injection, participants will return for an additional skin assessment of the treated areas.

DETAILED DESCRIPTION:
Objectives:

Our primary objectives are: to assess safety and tolerability of Intradermal electroporation (IDEP) using Derma Vax(Trademark) administered after pretreatment with either EMLA(Registered Trademark) cream as topical anesthetic or with placebo and to determine if the EMLA(Registered Trademark) cream applied to the electroporation site significantly decreases pain associated with the IDEP procedure. Our secondary objectives are: to determine the magnitude of pain perception of IDEP; to determine the quality of pain perception during IDEP using a Visual Analog Scale and the McGill pain scale; to determine the time course after IDEP of Pain rating and skin irritation and to determine variations in skin resistance with and without EMLA(Registered Trademark) cream and between participants.

Experimental Design and Methods:

Twelve healthy men or women will be recruited for this study. This is a randomized double-blind, placebo-controlled study with a medical device. Each subject will receive EMLA(Registered Trademark) cream or control cream placed on the electroporation site on each deltoid area in a blinded randomized manner. This will be followed by IDEP administration to each pre-treated deltoid area.

Medical Relevance and Expected Outcome:

DNA vaccines are a promising treatment for infectious diseases and cancer. The ideal delivery method for induction of cellular and humoral immune responses has not been defined. Information from this study is necessary for future studies using Derma Vax(Trademark) in therapeutic DNA vaccine studies. Derma Vax(Trademark) is unique in its proprieties of delivering a series of electric pulses that provoke DNA uptake by antigen presenting cells that reside in the dermal layer of the skin. We expect that the application of Intradermal Electroporation (IDEP) using Derma Vax(Trademark) will be well tolerated and the use of EMLA(Registered Trademark) cream will decrease the pain compared to placebo.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Female and male subjects, age 18 to 55 and in good health as determined by past medical history, physical examination, vital signs, electrocardiogram, and laboratory tests.
* Body mass index (BMI) must be within the range of 18 to 30 kg/m(2), inclusive
* Vital signs should be within the following ranges at screening and baseline:

  1. Oral body temperature between 35.0-37.5 degree C
  2. Systolic blood pressure, 85-140 mm Hg
  3. Diastolic blood pressure, 50-90 mm Hg
  4. Pulse rate, 50 - 100 bpm
* Ability to provide an informed consent.
* Blood tests demonstrating normal physiologic organ functions:

  1. Hematological (neutrophils greater than or equal to 1000; hemoglobin greater than or equal to 12 g/dl (female) and greater than or equal to 14g/dl (male); platelets > 150,000).
  2. Creatinine (Cre < 1.5 times ULN)
  3. LFTs (SGOT, SGPT, < 2.5 times ULN)
  4. PT and/or PTT < 1.5 times ULN

EXCLUSION CRITERIA:

* Participation in any clinical investigation within 4 weeks prior to dosing or longer if required by local regulations, and for any other limitation of participation based on local regulations.
* Significant illness within two weeks prior to dosing.
* History of clinically significant drug allergy or history of atopic allergy (asthma, urticaria, eczematous dermatitis)
* History of chronic skin disease that might interfere with IDEP application
* Known allergic reactions to adhesive tape
* History of use of chronic or current pain medication (narcotics)
* Sunburn or tattoos at the application sites (both shoulders)
* Subject has a pacemaker or implanted defibrillator
* A past medical history of clinically significant EKG abnormalities or a family history (grandparents, parents and siblings) of a sudden cardiac death or dysrhythmia.
* History of drug or alcohol abuse within the 12 months prior to dosing.
* History of noncompliance to medical regimens or unwillingness to comply with the study protocol
* History of HIV or hepatitis B or C.
* Pregnancy
* Known allergy to local anesthetics such as lidocaine

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2009-06-25; Primary Completion 2010-05-27 (Actual); Study Completion 2010-05-27 (Actual)

PRIMARY OUTCOMES:
Safety & Tolerability of Derma Vax
VAS with/without EMLA

SECONDARY OUTCOMES:
McGill Questionnaire and Present Pain Intensity with/without EMLA
Time course Visual Analogue Scale (VAS) and skin irritation and skin resistance

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Aging, Harbor Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Background] Lowe DB, Shearer MH, Kennedy RC. DNA vaccines: successes and limitations in cancer and infectious disease. J Cell Biochem. 2006 May 15;98(2):235-42. doi: 10.1002/jcb.20775. PMID 16440328
- [Background] Tang DC, DeVit M, Johnston SA. Genetic immunization is a simple method for eliciting an immune response. Nature. 1992 Mar 12;356(6365):152-4. doi: 10.1038/356152a0. PMID 1545867
- [Background] Srivastava IK, Liu MA. Gene vaccines. Ann Intern Med. 2003 Apr 1;138(7):550-9. doi: 10.7326/0003-4819-138-7-200304010-00011. PMID 12667025